CLINICAL TRIAL: NCT03176966
Title: Ropinirole for the Treatment of Muscle Cramps in Patients With Cirrhosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Andrew Scanga, Principal Investigator, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 160960
Record Dates: First submitted 2017-06-02; First posted 2017-06-06 (Actual); Results first posted 2022-10-31 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-09

CONDITIONS: Muscle Cramp; Cirrhosis
MeSH Terms: conditions — Muscle Cramp; Fibrosis | interventions — Vitamin E; ropinirole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vitamin E then Ropinirole (Active Comparator): Patients will be provided with vitamin E, 400 international units (IU), at baseline. Patient demographics will be collected along with baseline lab data including magnesium, potassium, albumin, and total bilirubin levels. After 3 months, patients will be switched to Ropinirole. Surveys measuring muscle cramp frequency and intensity will be collected at baseline, 3 months, and 6 months.
  Interventions: Drug: Vitamin E; Drug: Ropinirole; Other: Muscle cramp survey
- Ropinirole then Vitamin E (Active Comparator): Patients will be prescribed ropinirole at baseline. Patient demographics will be collected along with baseline lab data including magnesium, potassium, albumin, and total bilirubin levels. After 3 months, patients will be switched to vitamin E, 400 international units (IU). Surveys measuring muscle cramp frequency and intensity will be collected at baseline, 3 months, and 6 months.
  Interventions: Drug: Vitamin E; Drug: Ropinirole; Other: Muscle cramp survey

INTERVENTIONS:
Drug: Vitamin E — Patients will take 400 IU vitamin E nightly for 3 months.
Drug: Ropinirole — Patients will take 0.5mg ropinirole nightly for 3 months.
  Other Names: Requip
Other: Muscle cramp survey — Patients will complete a survey of muscle cramp frequency and severity at baseline, 3 months, and 6 months.

SUMMARY:
The investigator's aim is to compare the efficacy of Ropinirole (Requip) to vitamin E in the treatment of muscle cramps in cirrhotic patients.

DETAILED DESCRIPTION:
Muscle cramps are common in liver disease, especially in patients with cirrhosis. Despite the association of muscle cramps with liver disease, there is a paucity of information regarding treatment in these patients. Many treatment options have been reported in the literature but no standard of treatment has been established.

Oral vitamin E replacement has been used successfully in the management of nocturnal muscle cramps in cirrhotic patients. Ropinirole is primarily used for treatment of restless leg syndrome. An off label trial of low dose Ropinirole in clinical practice has shown some success in providing relief of muscle cramps in patients with cirrhosis. This study will compare Ropinirole to vitamin E treatment in a prospective cross-over study.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 18 years of age in the Vanderbilt Medical Center Hepatology Practice
* diagnosis of cirrhosis
* Self report regular muscle cramping

Exclusion Criteria:

* Patients without cirrhosis
* Patients under the age of 18
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2016-09-02 (Actual); Primary Completion 2021-10-22 (Actual); Study Completion 2021-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Scanga, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 31 subjects were consented and randomized. 1 subject became ill after randomization and was unable to participate so only 30 subjects took a first dose of assigned drug.
Period: Baseline to 3 Months (1st Intervention)
Arm/Group | Vitamin E Then Ropinirole | Ropinirole Then Vitamin E
Started | 14 | 16
Completed | 10 | 9
Not Completed | 4 | 7
Not completed — Death | 2 | 1
Not completed — Withdrawal by Subject | 1 | 4
Not completed — Lost to Follow-up | 1 | 2
Period: 3 Month to 6 Months (2nd Intervention)
Arm/Group | Vitamin E Then Ropinirole | Ropinirole Then Vitamin E
Started | 10 | 9
Completed | 4 | 4
Not Completed | 6 | 5
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 3 | 4
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Population: One subject was consented and randomized to Ropinirole then Vitamin E but became ill and withdrew prior to first dose of drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Vitamin E Then Ropinirole | Ropinirole Then Vitamin E | Total
Number analyzed (Participants) | 14 | 16 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.6 (8.8) | 61.8 (6.5) | 58.0 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 9 | 13
  Male | 10 | 7 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 14 | 14 | 28
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 14 | 14 | 28
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 14 | 16 | 30

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Muscle Cramps as Assessed by Patient Survey
Description: Compare the incidence of muscle cramps in patients using vitamin E versus ropinirole. Patients complete a survey that assesses the frequency of muscle cramps from once weekly or less to multiple episodes per day. Frequency scale is 0 to 3 with 0 being once weekly or less and 3 being multiple episodes a day. Survey is completed at the end of 3 months on study intervention.
Time Frame: 3 months
Population: Of the 23 participants who received Vitamin E, data was analyzed for those who completed the survey at the end of each specific crossover period (n=14). Of the 26 participants who received Ropinirole, data was analyzed for those who completed the survey at the end of each specific crossover period (n=13).
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Vitamin E Taken Nightly for 3 Months: Patients will be provided with vitamin E, 400 international units (IU), at baseline. Patient demographics will be collected along with baseline lab data including magnesium, potassium, albumin, and total bilirubin levels. .
  Vitamin E: Patients will take 400 IU vitamin E nightly for 3 months.
- Ropinirole Taken Nightly for 3 Months: Patients will be prescribed ropinirole at baseline. Patient demographics will be collected along with baseline lab data including magnesium, potassium, albumin, and total bilirubin levels.
  Ropinirole: Patients will take 0.5mg ropinirole nightly for 3 months.
Arm/Group | Vitamin E Taken Nightly for 3 Months | Ropinirole Taken Nightly for 3 Months
Number analyzed (Participants) | 14 | 13
score on a scale | 1.14 (0.99) | 1.23 (1.42)

2. Secondary Outcome: Muscle Cramp Severity as Assessed by Patient Survey
Description: Compare the severity of muscle cramps in patients using vitamin E versus ropinirole. Patients complete a survey that assesses muscle cramp pain on a scale from 0 to 10 with 0 being no pain and 10 being hurts worst. Survey is completed at the end of 3 months of study intervention.
Time Frame: 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vitamin E Taken Nightly for 3 Months | Ropinirole Taken Nightly for 3 Months
Number analyzed (Participants) | 14 | 13
score on a scale | 6.57 (3.79) | 6.00 (3.53)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for each patient while they remained on study for a maximum of 6 months participation.
Description: All cause mortality deaths were unrelated to any study intervention. These are not designated as SAEs.
Groups:
- Vitamin E: Patients will be provided with vitamin E, 400 international units (IU), at baseline. Patient demographics will be collected along with baseline lab data including magnesium, potassium, albumin, and total bilirubin levels. .
  Vitamin E: Patients will take 400 IU vitamin E nightly for 3 months.
- Ropinirole: Patients will be prescribed ropinirole at baseline. Patient demographics will be collected along with baseline lab data including magnesium, potassium, albumin, and total bilirubin levels.
  Ropinirole: Patients will take 0.5mg ropinirole nightly for 3 months.
Arm/Group | Vitamin E | Ropinirole
All-Cause Mortality (participants affected / at risk) | 3/23 | 1/26
Serious Adverse Events (participants affected / at risk) | 1/23 | 0/26
Other Adverse Events (participants affected / at risk) | 1/23 | 3/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vitamin E (N=23) | Ropinirole (N=26)
hepatic encephalopathy (Hepatobiliary disorders) | 1 (1) | 0 (0) — Subject admitted to hospital with altered mental status.Note suggests subject not compliant with prescribed lactulose. Subject discharged after one day. This event is not thought by the PI to be related to study IP or study related procedures.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vitamin E (N=23) | Ropinirole (N=26)
chest pressure (Cardiac disorders) | 0 (0) | 1 (1)
Increased muscle cramps (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nausea and vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
bruising (Blood and lymphatic system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-11): https://cdn.clinicaltrials.gov/large-docs/66/NCT03176966/Prot_SAP_000.pdf